CLINICAL TRIAL: NCT01151930
Title: Long-Term Compassionate Use Study for Continued Administration of SCB01A In Subjects Who Completed Treatment With SCB01A in the Previous Protocol # SCB01A-01
Brief Title: Long-Term Compassionate Use Study for Continued Administration of SCB01A-01
Status: No longer available | Type: Expanded Access
Sponsor: SynCore Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: SCB01A-01-B
Record Dates: First submitted 2010-06-23; First posted 2010-06-29 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2017-10

CONDITIONS: Malignant Solid Tumour
Keywords: Advanced solid tumor failed with standard therapy

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: SCB01A — This is a companion study to the protocol SCB01A-01 intended to provide long-term continued administration to subjects that completed Protocol SCB01A-01 on a compassionate basis. It is an open-label, single-arm study of SCB01A in subjects who have completed 2 cycles of treatment under the SCB01A-01 protocol.

SUMMARY:
The primary objective is to characterize the safety profile of long-term exposure to SCB01A when administered to cancer subjects with advanced solid tumors. Furthermore, the efficacy profile will also be explored in this study.

DETAILED DESCRIPTION:
This is a companion study to the protocol SCB01A-01 intended to provide long-term continued administration to subjects that completed Protocol SCB01A-01 on a compassionate basis. It is an open-label, single-arm study of SCB01A in subjects who have completed at least one cycles of treatment under the SCB01A-01 protocol.

ELIGIBILITY:
Inclusion Criteria:

Subjects who completed protocol SCB01A-01 and exhibited a favorable response or had no clinical evidence of disease progression (i.e. stable disease, partial response or complete response).

Exclusion Criteria:

Study participants meeting any of the following criteria will be excluded from enrollment:

1. Unwilling or unable to provide informed consent.
2. Unwilling or unable to comply with the requirements of the protocol.
3. Has unresolved toxicities from previous SCB01A-01 protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

REFERENCES:
- [Derived] Shiah HS, Chiang NJ, Lin CC, Yen CJ, Tsai HJ, Wu SY, Su WC, Chang KY, Wang CC, Chang JY, Chen LT. Phase I Dose-Escalation Study of SCB01A, a Microtubule Inhibitor with Vascular Disrupting Activity, in Patients with Advanced Solid Tumors. Oncologist. 2021 Apr;26(4):e567-e579. doi: 10.1002/onco.13612. Epub 2020 Dec 18. PMID 33245172